CLINICAL TRIAL: NCT01860599
Title: The Effect of Controlled Aerobic Exercise on Endothelial Dysfunction and Vascular Reactivity in Patients With Pre-diabetes: A Crossover Pilot Study
Brief Title: Effects of Aerobic Exercise in Patients With Pre-diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baystate Medical Center (Other)
Responsible Party: Principal Investigator, Sabyasachi Sen, MD, Assistant Professor Endocrinology, Baystate Medical Center
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: IRB132171
Record Dates: First submitted 2013-05-09; First posted 2013-05-23 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Prediabetes
Keywords: prediabetes; EPC's; vascular reactivity
MeSH Terms: conditions — Prediabetic State | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Prediabetes with exercise (Other): 150 minutes of moderate exercise per week
  Interventions: Behavioral: Exercise
- Prediabetes without exercise (Other): Pre-study activity level (i.e. no exercise)
  Interventions: Behavioral: Without exercise

INTERVENTIONS:
Behavioral: Exercise — 150 minutes of moderate exercise per week
  Arms: Prediabetes with exercise
Behavioral: Without exercise — Pre-study activity level (i.e. no exercise)
  Arms: Prediabetes without exercise

SUMMARY:
It is well known that diabetes and excessive or high blood sugars causes blood vessel and blood cell damage. It is also possible, then, that people with pre-diabetes may also start to have blood vessel and blood cell damage as the blood sugars rise from the normal range into the diabetic range. In addition to looking at potential damage, the question is whether or not this damage improves with exercise. This study aims to look at blood vessel and blood cells in three different ways by 1) looking at how the blood vessel responds to "sheer force" (a blood pressure cuff pumped up and then released after a few minutes). This is done by ultrasound. 2) By looking at blood tests such as blood sugar, cholesterol, and inflammation and 3) By looking at certain blood cells in the lab, how long they live and the number of cells left after a certain number of days, and again, if this improves with exercise.

DETAILED DESCRIPTION:
* To refine a non-invasive test for endothelial dysfunction. The investigators will examine the flow response to sheer-stress induced by the relief of pressure exerted with a blood pressure cuff on the brachial artery, measuring flow responses with Doppler. This is a measure of local nitric oxide production from endothelial cells which is known to be impaired in diabetics, normal in non-diabetics, but unknown in prediabetics.
* To measure in the same individuals indicators of glucose metabolism abnormalities including fasting blood glucose, HbA1C, insulin sensitivity by homeostasis model assessment-estimated insulin resistance (HOMA-IR) and insulin levels.
* To measure Endothelial Progenitor Cell (EPC) count, viability, gene expression of key genes such as endothelial nitric oxide synthase (eNOS), von-Willebrand's Factor (vWF) and adhesion molecules such platelet-endothelial cell adhesion molecule-1 (PECAM-1 or CD31), cadherin such as Vascular-Endothelial cadherin (VE-cadherin)or CD (cell surface marker)-144, growth factors such as vascular-endothelial growth factor (VEGF)and Insulin like growth factor (IGF-1)in the EPCs from pre-diabetes subjects pre and post exercise.
* Correlate the glucose metabolism abnormalities with potential causative factors of endothelial dysfunction by studying EPC functions such as migration and tube formation and susceptibility to apoptosis in moderate hyperglycemia. Apoptosis assay will be done by Flow Cytometry analysis using Annexin V- Propidium-iodide dye.
* Subjects will be randomized to the intervention (structured exercise) or continuation of their usual life style (non-exercise, sedentary)group.

In both arms of the study, subjects will be encouraged to adhere to the standard dietary advice that all pre-diabetic patients receive as part of their standards of care, irrespective of design arm they will be in.

The investigators expect exercise to improve flow-mediated vasodilatation, EPC colony count and function, along with better key gene expressions noted by Real Time-qualitative polymerase chain reaction (PCR).

* Assess the effects of the intervention comparing them to the findings in each individual, in a paired manner.
* After a washout period, individuals will be crossed over to see whether the effects of the intervention are reversed and to demonstrate that the difference between controls and intervention subjects was due to the aerobic exercise intervention, and not due to random differences

ELIGIBILITY:
Inclusion Criteria:

* Prediabetic

  * Impaired fasting glucose (100-125mg/dl)
  * Impaired glucose tolerance (2' post between 140-199mg/dl)
  * HbA1C 5.7-6.4 mg/d (inclusive)
* Exercise Naive
* BMI between 20-39.9
* Nutritional Counseling prior to participation with CDE/RD
* Willing to wear activity monitor
* Willing to keep a dietary log

Exclusion Criteria:

* Pace maker or other implanted device that might have interference with Tanita scale
* Any contraindication to moderate exercise
* Previous coronary disease or cerebrovascular event active or clinically significant coronary vascular disease, or peripheral vascular disease
* Diabetes
* Uncontrolled hypertension (SBP > 140 or DBP > 90 on 3 separate occasions) ACE's or ARB's
* Premature familial CAD (Father < 55years____ Mother <65years)
* HDL < 40mg/dl
* Triglycerides >400mg/dl
* Any new lipid lowering medication started in the past 6 months
* Framingham Risk Score two or more

  1. Smoking
  2. Hypertension (B/P > 140/90 or on antihypertensives)
  3. HDL < 40mg/dl
  4. Age men >45years or women >55years
* Low hematocrit ( or hemoglobinopathies that may impair exercise tolerance) or abnormal CBC
* Uncontrolled hypo/hyperthyroidism
* Active smoking
* Liver disease ( alt or AST> 2.5's UNL)
* Moderate or Severe Kidney disease, current or history
* Pancreatitis, current or history
* Any medication started in the last 3 months
* Active non healing wounds
* Recent Surgery in the last 3 months
* Anti-inflammatory disease, current or history
* Regular use of anti-inflammatory drugs
* CA
* Alcoholism
* Women who are pregnant or intending to become pregnant
* Oral or Injectable antidiabetic medication
* Post menopausal women on hormone replacement
* Any steroid medication (oral, inhaled, injected or nasal)

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-03; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Measures of Endothelial Function by studying number, function and gene expression of endothelial progenitor cells (identified as CD34+ cells) | 16 weeks per patient
  A. Number of viable CD34 +ve cells at Day-0 and viability assay. B. Colony Formation count assay at Day-5, pre and post exercise. C. We will test CD34+ cell migration, adhesion and tube formation properties. D. Gene expression in CD34+ cells of critical endothelial function and inflammatory genes will be measured: eNOS, vWF and PECAM1, VE-cadherin, VEGF-A, Superoxide dismutase (SOD)-1, 2 and 3, Catalase, Interleukin (IL)-6, Tumor Necrosis Factor (TNF alpha), P53, P21, PUMA, Bcl2 [Apoptosis genes] will also be noted

SECONDARY OUTCOMES:
Measures of Vacular Reactivity | 16 weeks
  A) Measure Brachial reactivity through shear-stress using flow mediated dilatation (FMD) B). Measure Arterial Stiffness measure pre and post exercise. C) Measure Carotid Intima Media Thickness will be measured at each time point

OTHER OUTCOMES:
Measures of Insulin Sensitivity by measuring inflammatory molecules as a surrogate of insulin resistance | 16 weeks
  We will measure:
  A. plasma measurements of cytokines, including C - reactive protein, E-selectin, IL-6, IL-10, thrombin, leptin, adiponectin, fasting glucose, fasting insulin and fasting lipid profile from subjects are expected to reflect endothelial inflammation.
  B. Insulin sensitivity will be evaluated at baseline and weeks 6, 10 and16 using the HOMA ratio, calculated from individual serum measures (fasting glucose* insulin/405) C.Adiposity will be measured at baseline and at weeks 6, 10, and 16 using the Tanita Body Composition Analyzer scale, measured as percentage body fat D. Resting energy expenditure as measures of indirect calorimetry for basal metabolic rate measures (BMR).

CONTACTS AND LOCATIONS:
Overall Officials: Sabyasachi Sen, MD, PhD, Principal Investigator — Baystate Medical Center
Locations (1):
- Baystate Medical Center, Springfield, Massachusetts, United States